CLINICAL TRIAL: NCT05853575
Title: A Randomized Study of Two Dosing Regimens of Adagrasib in Patients With Previously Treated Non-Small Cell Lung Cancer With KRAS G12C Mutation
Brief Title: Trial of Two Adagrasib Dosing Regimens in NSCLC With KRAS G12C Mutation (KRYSTAL 21)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA239-0012; 2023-503523-25 (Other: EU CT Number); CA239-0012 (Other: Bristol-Myers Squibb Protocol ID); 849-021 (Other: Mirati Therapeutics Protocol ID)
Expanded Access: NCT05162443 (Approved for marketing)
Record Dates: First submitted 2023-04-12; First posted 2023-05-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Advanced Cancer; Metastatic Cancer; Malignant Neoplasm of Lung
Keywords: KRAS G12C; Non-small cell lung cancer; Metastatic cancer; NSCLC
MeSH Terms: conditions — Neoplasm Metastasis; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adagrasib 600mg BID (Experimental): Adagrasib 600mg BID without regard to food
  Interventions: Drug: Adagrasib
- Adagrasib 400mg BID (Experimental): Adagrasib 400mg BID with food
  Interventions: Drug: Adagrasib

INTERVENTIONS:
Drug: Adagrasib — KRAS G12C inhibitor
  Other Names: MRTX849; Krazati

SUMMARY:
This study will evaluate the efficacy of two dosing regimens of adagrasib (600 mg BID versus 400 mg BID) in patients with NSCLC with KRAS G12C mutation.

DETAILED DESCRIPTION:
CA239-0012 is a phase 2 study of adagrasib monotherapy in which patients are randomized between two dosing regimens. The study will evaluate the efficacy of two dosing regimens of adagrasib (600 mg BID without regard to food versus 400 mg BID with food) in patients with NSCLC with KRAS G12C mutation and who have received prior treatment with a platinum-based regimen and immune checkpoint inhibitor therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Are at least 18 years old (or old enough to legally make their own treatment decisions, according to local laws).
* Have advanced NSCLC or metastatic NSCLC (NSCLC that started in the lungs and then spread to other parts of the body) with the KRAS G12C mutation.
* Have had previous treatment with 1) chemotherapy that included a drug called cisplatin or a drug called carboplatin and 2) a type of drug called an immune checkpoint inhibitor.
* Have recovered from their prior treatment and blood tests are within a safe range.

Key Exclusion Criteria:

* Have had previous treatment with a drug that targets KRAS G12C.
* Have cancer that can potentially be removed with surgery.
* Patients with brain lesions are not eligible if 1) any untreated brain lesions are > 2.0 cm in size 2) any brainstem lesions are present 3) ongoing steroid dosing >10 mg daily prednisone (or equivalent) and 4) poorly controlled (> 1/week) generalized or complex partial seizures or neurologic progression/instability due to brain lesions.
* Have certain medical conditions or need to take certain medications that, in the opinion of a trial doctor, could make it unsafe for them to participate or difficult to complete the trial assessments, or are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). | 30 months
  ORR evaluation of subjects treated with adagrasib 600 mg BID without regard to food versus 400 mg BID with food having NSCLC with KRAS G12C mutation (Study Population) will be completed per blinded independent central radiology (BICR) review. Objective response is the proportion of subjects that experience confirmed complete response (CR) or partial response (PR) based on RECIST v1.1 during the time period from 1st dose of adagrasib until last dose of adagrasib.

SECONDARY OUTCOMES:
Evaluate Overall Survival (OS). | 45 months
  Overall survival is defined as time from date of randomization to date of death due to any cause.
Evaluate Progression Free Survival (PFS). | 30 months
  Progression-free survival is defined as time from date of randomization to date of first progression per RECIST 1.1 or death from any cause, whichever occurs first.
Evaluate Duration of Response (DOR). | 30 months
  Duration of response defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of either PD (per BICR review) or death due to any cause, whichever occurs first.
Safety and tolerability in the study population. | 30 months
  Safety characterized by number of participants with AEs, with abnormal laboratory test results and number of patients modifying or discontinuing study treatment due to an AE:
  1. Type, incidence, severity, timing, seriousness, and relationship to study treatment of Adverse Events.
  2. Laboratory abnormalities as measured by changes in lab results such as hematologic or chemistry parameters while on study treatment.
  3. Number of patients modifying or discontinuing study treatment due to Adverse Event.
Population pharmacokinetic (PK) Model Derived Area Under the Curve During the Dosing Interval at Steady State (AUCtau,ss). | Pre-dose and 4-6 hours post dose; up to 6 months.
  Sparse concentration data from this study will be pooled with other studies and analyzed using population PK methods to derive individual exposure parameters. Data for this Outcome Measure will not be reported here since ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Patient-reported symptoms during adagrasib administration from first dose to 28 days after last dose of adagrasib. | 30 months
  Patient reported outcomes (PROs) will be used to assess symptomatic toxicity of adagrasib using the NCI Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Measurement System. PRO items reflect the specific symptom 1) frequency, severity, interference with usual or daily activities, 2) amount, or 3) presence or absence. PRO-CTCAE responses are scored from 0 (low) to 4 (high), or 0/1 for absent/present, and scores for each attribute (frequency, severity and/or interference) are presented descriptively.
Patient -reported quality of life during adagrasib administration from first dose to End of Treatment visit. | 30 months
  Patient reported quality of life questionnaire will be used to assess five dimensions of patient health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using the 5-Level EQ-5D version (EQ-5D-5L) established by the EuroQol Group. This is presented descriptively, and patient responses correspond to a value of 1 (low) or 5 (high). Additionally, a one- page Visual Analog Scale (VAS) will be provided to patients so they may report their self-rated health from the best (100) and worst (0) health imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (118):
- United States (6):
  - Local Institution - 101, Santa Rosa, California
  - Local Institution - 104, Chicago, Illinois
  - Local Institution - 103, Minneapolis, Minnesota
  - Kansas City VA Hospital, Kansas City, Missouri
  - Veterans Affairs Medical Center (VAMC) - Durham - Oncology, Durham, North Carolina
  - VA North Texas Healthcare System/Dallas VA Medical Center, Dallas, Texas
- Brazil (5):
  - Ensino e Terapia de Inovação Clinica AMO-ÉTICA / Ética Pesquisa e Ensino, Salvador, Estado de Bahia
  - Uniao Brasileira de Educacao E Assistencia, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Oncocentro Belo Horizonte, Belo Horizonte, São Paulo
  - A.C. Camargo Cancer Center, São Paulo
- Croatia (3):
  - Klinički bolnički centar Sestre milosrdnice, Zagreb, City of Zagreb
  - Local Institution - 525, Pula, Istria County
  - Specijalna Bolnica Medico - Rijeka, Rijeka, Primorje-Gorski Kotar County
- France (13):
  - CHU de Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - Hopital Haut-Leveque - Maladies respiratoires, Pessac, Gironde
  - Institut de Cancerologie de I'Ouest - Service d'Oncologie Medicale - Service d'Oncologie Médicale, Saint-Herblain, Loire-Atlantique
  - Centre Hospitalier Universitaire D' Angers Hôpital Larrey - PNEUMOLOGIE - Département de PNEUMOLOGIE, Angers, Maine-et-Loire
  - CHU de Nantes - HÃ´pital Nord LaÃ"nnec (HGRL) - Service dOncologie medicale â€" Unite dOncologie thoracique, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Poitiers - Service d'oncologie Médicale Oncologie Medicale - Cancerolo, Poitiers, Poitou-Charentes
  - Centre Hospitalier Universitaire de Nice, Nice, Provence-Alpes-Côte d'Azur Region
  - AP-HM Hopital Nord, Marseille, Rhône
  - Centre Hosptalier De Villefranche-Sur-Saone - Oncologie Medicale - Cancerolo, Villefranche-sur-Saône, Rhône
  - Centre Hôspitalier de Bretagne Sud - Hôpital du Scorff, Lorient
  - GIE Groupe hospitalier Paris Saint-Joseph/Vinci, Paris
  - Centre Hospitalier de Cornouaille, Quimper
  - Hôpital Bégin - Service d'Oncologie, Saint-Mandé
- Greece (7):
  - Local Institution - 577, Pátrai, Achaïa
  - General Hospital of Athens "Alexandra", Athens, Attica
  - Local Institution - 582, Athens, Attica
  - Attikon Hospital - 2nd Critical Care, Haidari - Athens, Pella
  - St. Luke's Hospital S.A., Panórama
  - Theageneio Cancer Hospital, Thessaloniki
  - General Hospital Of Thessaloniki Papageorgiou, Thessaloniki
- Hungary (2):
  - Local Institution - 600, Szolnok, Jász-Nagykun-Szolnok
  - Local Institution - 603, Debrecen
- Israel (5):
  - Shaare Zedek Medical center, Jerusalem, Jerusalem
  - Bnai Zion Medical Center Rheumatology Unit, Haifa, Tel Aviv
  - Assuta Medical Center, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus, Haifa
  - Tel Aviv Sourasky Medical Center - Oncology - Hematology/Oncology, Tel Aviv
- Italy (6):
  - Azienda Sanitaria Territoriale Pesaro Urbino (AST PU), Pesaro, Pesaro E Urbino
  - Azienda Ospedaliero-Universitaria Maggiore Della Carita, Novara, Piedmont
  - Istituto di Candiolo, IRCCS, Candiolo, Torino
  - IEO - Istituto Europeo di Oncologia, IRCCS, Milan
  - Ospedale S.Maria della Misericordia, AO di Perugia, Università degli Studi di Perugia, Perugia
  - Istituto Nazionale Tumori Regina Elena - IRCCS - IFO, Roma
- Japan (4):
  - Ehime University Hospital, Tōon, Ehime
  - Local Institution - 403, Nishinomiya, Hyôgo [Hyogo]
  - National Cancer Center Hospital East, Kashiwa, Tiba [Chiba]
  - Local Institution - 400, Osaka, Ôsaka [Osaka]
- Mexico (4):
  - Local Institution - 128, Tuxtla Gutiérrez, Chiapas
  - Local Institution - 129, Colonia Nápoles, Mexico City
  - Local Institution - 127, Colonia Roma, Mexico City
  - Local Institution - 125, Toluca
- Netherlands (3):
  - Local Institution - 802, Breda, North Brabant
  - Anthoni van Leeuwenhoek Ziekenhuis, Nederlands Kanker Instit, Amsterdam, North Holland
  - St. Antonius Hospital, Utrecht
- Peru (2):
  - Local Institution - 152, San Martín de Porres, Lima region
  - Local Institution - 151, Surquillo, Lima region
- Poland (3):
  - Local Institution - 650, Krakow, Lesser Poland Voivodeship
  - Local Institution - 651, Gdynia, Pomeranian Voivodeship
  - Local Institution - 653, Lublin
- Romania (10):
  - Medisprof - Medical Oncology, Cluj-Napoca, Cluj
  - Ovidius Clinical Hospital, Ovidiu, Constanța County
  - Local Institution - 727, Craiova, Dolj
  - Oncolab - Medical Oncology, Craiova, Dolj
  - Centrul de Oncologie Sf Nectarie - Medical Oncology, Craiova, Dolj
  - Oncocenter- Oncologie Clinica - Medical Oncology, Timișoara, Timiș County
  - Local Institution - 726, Bucharest
  - Centrul de Oncologie Euroclinic, Iași
  - Spitalul Clinic Judetean De Urgenta Sibiu, Sibiu
  - Sigmedical Services S.R.L., Suceava
- Serbia (5):
  - Local Institution - 750, Kamenitz, Vojvodina
  - University Clinical Center of Nis, Clinic for Pediatrics-Department for Pulmonology, Nis, Vojvodina
  - Local Institution - 753, Belgrade
  - Local Institution - 751, Belgrade
  - University Clinical Center of Kragujevac, Center for Internal Oncology, Kragujevac, Šumadijski Okrug
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggido [Kyonggi-do]
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Local Institution - 328, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Local Institution - 326, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
- Spain (15):
  - Complejo Hospitalario Universitario De Santiago - Oncología Médica, Santiago de Compostela, A Coruña
  - Hospital Regional Universitario De Málaga, Málaga, Andalusia
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Local Institution - 686, Santander, Cantabria
  - Local Institution - 676, Oviedo, Principality of Asturias
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Dexeus Grupo Quironsalud, Barcelona
  - Hospital Universitario Vall d'Hebron - Oncología Médica, Barcelona
  - Local Institution - 689, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Local Institution - 679, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Virgen de la Macarena - Oncología Médica, Seville
  - Hospital Clinico Universitario De Valencia - Oncologia Médica y Hematologia, Valencia
  - Local Institution - 684, Valencia
- Taiwan (6):
  - Local Institution - 351, Kaohsiung City, Kaohsiung
  - Chang Gung Medical Foundation - Kaohsiung Chang Gung Memorial Hospital, Kaohsuing City, Kaohsiung
  - Chung Shan Medical University Hospital - Internal Medicine, Taichung, Taichung
  - China Medical University Hospital - Internal Medicine, Taichung, Taichung
  - Local Institution - 355, Taichung, Taichung
  - Local Institution - 354, Taipei City, Taipei
- Thailand (4):
  - Local Institution - 376, Muang, Chiang Mai
  - Local Institution - 377, Bangkok, Krung Thep Maha Nakhon [Bangko
  - Local Institution - 375, Khon Kaen
  - Holistic Center for Cancer Study and Care, Songkhla
- Turkey (Türkiye) (11):
  - Memorial Ankara Hastanesi, Ankara, Ankara/Cankaya
  - Gülhane Eğitim ve Araştırma Hastanesi, Ankara, Etlik/Ankara
  - Medipol Mega Hospital, Istanbul, Samsun
  - Istanbul Oncology Hospital - Medical Oncology, Istanbul, Samsun
  - Local Institution - 703, Istanbul, Samsun
  - Dr Abdurrahman Yurtaslan Training and Research Hospital - Medical Oncology, Ankara
  - Ankara Liv Hospital, Ankara
  - Ankara City Hospital - Medical Oncology, Ankara
  - Trakya Univ Hastanesi Ic Hastal, Edirne
  - Goztepe SuleymanYalcin Sehir Hast, Istanbul
  - Ege University Medical Faculty - Pulmonary, Izmir

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05853575.html